CLINICAL TRIAL: NCT06428630
Title: Systemic Absorption of Dexamethasone Oral Rinse in Patients With Oral Lichen Planus
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study protocol changed to be a retrospective exempt review project.
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004549
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Oral Lichen Planus; Oral Lichenoid Reaction
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Intervention Model Description: Investigative group: Subjects with symptomatic oral lichen planus (OLP) or oral lichenoid reactions (OLR) Control Group: Those otherwise healthy
  Both groups will receive the same intervention. 5 of the control subjects will swish for 5 minutes, 5 of the control subjects will swish for 2 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Investigative group- Those with OLP (Experimental): The investigative will apply the dexamethasone oral rinse 0.5 mg/5ml treatment. The oral rinse is considered a topical rinse because it is confined to the oral cavity (topical) and not swallowed. Subjects will be reminded by the study team via a phone call a few days before their visit that they must not drink water or eat at least 60 min before their visit. Once we get to the stage of the rinse, we will first their oral cavity with gauze. Then, we will instruct the subject to Rinse their mouth with 0.5mg/5ml dexamethasone for 2 min, then spit into a provided plastic cup the oral rinse. This will then be discarded down the drain.
  Interventions: Drug: dexamethasone oral rinse
- Control 1 - 5 minute rinse (Active Comparator): The first control group will apply the dexamethasone oral rinse 0.5 mg/5ml treatment. The oral rinse is considered a topical rinse because it is confined to the oral cavity (topical) and not swallowed. Subjects will be reminded by the study team via a phone call a few days before their visit that they must not drink water or eat at least 60 min before their visit. Once we get to the stage of the rinse, we will first their oral cavity with gauze. Then, we will instruct the subject to Rinse their mouth with 0.5mg/5ml dexamethasone for 5 min, then spit into a provided plastic cup the oral rinse. This will then be discarded down the drain.
  Interventions: Drug: dexamethasone oral rinse
- Control 2- 2 minute rinse (Active Comparator): The second control group will apply the dexamethasone oral rinse 0.5 mg/5ml treatment. The oral rinse is considered a topical rinse because it is confined to the oral cavity (topical) and not swallowed. Subjects will be reminded by the study team via a phone call a few days before their visit that they must not drink water or eat at least 60 min before their visit. Once we get to the stage of the rinse, we will first their oral cavity with gauze. Then, we will instruct the subject to Rinse their mouth with 0.5mg/5ml dexamethasone for 2 min, then spit into a provided plastic cup the oral rinse. This will then be discarded down the drain.
  Interventions: Drug: dexamethasone oral rinse

INTERVENTIONS:
Drug: dexamethasone oral rinse — The study drug is FDA approved (NDC- 0054-3177) and will be used as it would be used in a standard of care setting. The rinse will be administered on the same therapeutic dose to OLP/OLR (0.5 mg/5ml of dexamethasone oral rinse once (rinse for 2 minutes or 5 minutes), then spit the excess into a cup.
  The oral rinse dexamethasone 0.5 mg/5ml will be used only on the subjects who participated in the study.

SUMMARY:
The objective of this study is to see the amount of systemic absorption of a standard dose of dexamethasone oral rinse for patients with symptomatic oral lichen planus (OLP) or oral lichenoid reactions (OLR) and healthy subjects (those who do not have OLP or OLR aka the control group).

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. Non-pregnant
3. Newly diagnosed subjects with OLP/OLR. Definition of 'newly" in this case : new patient with complaint regarding oral erosions and ulceration, and diagnose clinically with OLP or OLR for the first time
4. Those not exposed to topical or systemic corticosteroids for the previous 1 month. Meaning, those willing to not take this OLP/OLR treatment for 1 month before their visit
5. Experimental group is clinically diagnosed with OLP/OLR
6. Controls must have no history of OLP/OLR

Exclusion Criteria:

1 . Under 18 years old 2. Pregnant women 3. Recent history (< than one month) of exposure to topical or systemic corticosteroids.

4. History of advanced kidney, liver disease, or systemic fungal infection. 5. Corticosteroids hypersensitivity. 6. Active oral candidiasis 7. Patients on blood thinners medication ,anemic or suffer from bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Systemic absorption of a standard dose of dexamethasone oral rinse | 2 hours per subject
  To investigate the amount (level detected in blood), through blood draw, of how much dexamethasone oral rinse is absorbed in the blood stream over two hours.

SECONDARY OUTCOMES:
Assessment of correlation between the amount of systemic absorption and the severity of the oral mucosal disorder | 2 hours per subject
  A clinical oral examination will be conducted for the REU scoring system this will determine what severity category they are in (what their REU score is out of 30 with 30 being most severe and 0 being mild lichen planus). The oral cavity will be examined based on REU scoring system to determine the subject belong to mild , moderate or severe group.

OTHER OUTCOMES:
Length of rinsing impact on systemic absorption | 2 hours per subject
  If there is systemic absorption, does it differ based on length of time of rinsing? This is for those in the control group who will be rinsing for either 2 minutes or 5 minutes. The evaluation is if there is varying amounts of the rinse detected in the blood after the various blood draws.

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Sankar, DMD, MHS, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rice JB, White AG, Scarpati LM, Wan G, Nelson WW. Long-term Systemic Corticosteroid Exposure: A Systematic Literature Review. Clin Ther. 2017 Nov;39(11):2216-2229. doi: 10.1016/j.clinthera.2017.09.011. Epub 2017 Oct 19. PMID 29055500
- [Background] Meikle AW, Lagerquist LG, Tyler FH. A plasma dexamethasone radioimmunoassay. Steroids. 1973 Aug;22(2):193-202. doi: 10.1016/0039-128x(73)90085-8. No abstract available. PMID 4795381
- [Background] Spoorenberg SM, Deneer VH, Grutters JC, Pulles AE, Voorn GP, Rijkers GT, Bos WJ, van de Garde EM. Pharmacokinetics of oral vs. intravenous dexamethasone in patients hospitalized with community-acquired pneumonia. Br J Clin Pharmacol. 2014 Jul;78(1):78-83. doi: 10.1111/bcp.12295. PMID 24400953
- [Background] Jarvinen A, Granander M, Laine T, Viitanen A. Effect of dose on the absorption of estradiol from a transdermal gel. Maturitas. 2000 Apr 28;35(1):51-6. doi: 10.1016/s0378-5122(00)00101-8. PMID 10802400
- [Background] Aalto-Korte K, Turpeinen M. Quantifying systemic absorption of topical hydrocortisone in erythroderma. Br J Dermatol. 1995 Sep;133(3):403-8. doi: 10.1111/j.1365-2133.1995.tb02668.x. PMID 8546995
- [Background] Georgaki M, Piperi E, Theofilou VI, Pettas E, Stoufi E, Nikitakis NG. A randomized clinical trial of topical dexamethasone vs. cyclosporine treatment for oral lichen planus. Med Oral Patol Oral Cir Bucal. 2022 Mar 1;27(2):e113-e124. doi: 10.4317/medoral.25040. PMID 34564686
- [Background] Joly P, Roujeau JC, Benichou J, Picard C, Dreno B, Delaporte E, Vaillant L, D'Incan M, Plantin P, Bedane C, Young P, Bernard P; Bullous Diseases French Study Group. A comparison of oral and topical corticosteroids in patients with bullous pemphigoid. N Engl J Med. 2002 Jan 31;346(5):321-7. doi: 10.1056/NEJMoa011592. PMID 11821508
- [Background] Varoni EM, Molteni A, Sardella A, Carrassi A, Di Candia D, Gigli F, Lodi F, Lodi G. Pharmacokinetics study about topical clobetasol on oral mucosa. J Oral Pathol Med. 2012 Mar;41(3):255-60. doi: 10.1111/j.1600-0714.2011.01087.x. Epub 2011 Sep 22. PMID 21950548
- [Background] Sankar V, Hearnden V, Hull K, Juras DV, Greenberg MS, Kerr AR, Lockhart PB, Patton LL, Porter S, Thornhill M. Local drug delivery for oral mucosal diseases: challenges and opportunities. Oral Dis. 2011 Apr;17 Suppl 1:73-84. doi: 10.1111/j.1601-0825.2011.01793.x. PMID 21382140
- [Background] Plemons JM, Rees TD, Zachariah NY. Absorption of a topical steroid and evaluation of adrenal suppression in patients with erosive lichen planus. Oral Surg Oral Med Oral Pathol. 1990 Jun;69(6):688-93. doi: 10.1016/0030-4220(90)90349-w. PMID 2356081
- [Background] Einarsdottir MJ, Bankvall M, Robledo-Sierra J, Rodstrom PO, Bergthorsdottir R, Trimpou P, Hasseus B, Ragnarsson O. Topical clobetasol treatment for oral lichen planus can cause adrenal insufficiency. Oral Dis. 2024 Apr;30(3):1304-1312. doi: 10.1111/odi.14588. Epub 2023 Apr 27. PMID 37103329